CLINICAL TRIAL: NCT04091594
Title: Investigating the Effects of Sensory Input Orthotics in Disorders of Posture and Movement
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient funding was available and the study could not be started.
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: HM20015260
Record Dates: First submitted 2019-09-13; First posted 2019-09-17 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Flexible orthotic (Experimental): Sensory input flexible ankle foot orthotic (SIAFO) with appropriate lycra garments
  Interventions: Device: Flexible orthotic
- Standard of care (Active Comparator): Standard of care solid ankle foot orthotic (AFO)
  Interventions: Device: Standard orthotic

INTERVENTIONS:
Device: Flexible orthotic — Participants will receive the SIAFO to wear
  Arms: Flexible orthotic
Device: Standard orthotic — Participants will received the standard AFO to wear
  Arms: Standard of care

SUMMARY:
The purpose of this research study is to use tools for measuring function and movement in pediatric populations to measure the impact of input orthotic interventions in children with cerebral palsy.

DETAILED DESCRIPTION:
Sensory processing begets movement. In persons with disorders of posture and movement due to cerebral palsy, an impaired ability to integrate multiple senses including pressure from ground, limb proprioception, and vestibular inputs leads to a movement pattern that is coarse, spastic and inefficient. In the pediatric rehab clinic spastic movement disorders have been treated with flexible, molded orthotics for the foot and ankle (AFO) to enhance sensation of ground reaction forces, and flexible elastomeric compression garments to enhance body and limb proprioception. While the investigators observed substantial improvements in gait quality and postural stability using sensory input orthotics, these clinical observations have not been objectively quantified. The goal is to use validated tools for measuring function and movement in pediatric populations in order to gather data on the value of sensory input orthotic interventions in children with cerebral palsy.

Under the term, sensory input orthotic, the following items are included which will be used in this study. 1) A flexible, thin polypropylene shell ankle-foot orthotic designed according to Hylton et al. Journal of P&O 1989. 2) Wearable elastomeric compression garments manufactured by SPIO or from the Boston Brace DMO garment line. 3) A vibrating anklet that provides subsensory vibrational stimulation to the leg, manufactured by Accelera.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cerebral palsy
* Ages 6 months to 21 years
* No prior prescription of sensory input ankle-foot orthotics
* Clinical diagnosis of abnormal gait and mobility

Exclusion Criteria:

• Joint contracture that severely limits function such as ability to passively open the hand, extend the arm at the elbow or to stand with feet flat on the ground or knees in an extended position.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Change in perceived psychosocial well-being - parents | Baseline to 2 months
  Participant's parents will complete the Pediatric Evaluation of Disabilities Inventory (PEDI)
Change in perceived psychosocial well-being - children | Baseline to 2 months
  Children ages 9 and up will be administered the Psychosocial Impact of Assistive Device Survey (PIADS) by a trained clinician
Change in gross motor function | Baseline to 2 months
  A trained physical therapist will administer the global gross motor function (GMFM-88) assessment
Change in lower extremity kinematics and posture stability | Baseline to 2 months
  Participants will perform a 10 second walk test in the Motor Control Lab while being recorded with a Vicon 3D motion capture system.
Change in balance | Baseline to 2 months
  Participants will perform the 14-point items of the Pediatric Balance Scale in the Motor Control Lab while being recorded with a Vicon 3D motion capture system.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Rolin, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No